CLINICAL TRIAL: NCT02017795
Title: Managing Asthma With Tele-health Technology: A Feasibility Study
Brief Title: Asthma Self-management Via Application of Telehealth
Acronym: asthma
Status: Unknown | Phase: Not Applicable | Type: Interventional
Last Known Status: Active, not recruiting
Sponsor: University of British Columbia (Other)
Collaborators: Pfizer (Industry); Providence Health & Services (Other)
Responsible Party: Sponsor
Allocation: Randomized | Model: Parallel | Masking: Double | Purpose: Supportive Care
Other Study IDs: H13-02666
Record Dates: First submitted 2013-11-29; First posted 2013-12-23 (Estimated); Last update posted 2016-05-27 (Estimated); Status verified 2016-05

CONDITIONS: Asthma; Mixed Asthma With Acute Exacerbation
Keywords: asthma, mixed asthma, telehealth, action plan, exacerbation
MeSH Terms: conditions — Asthma

STUDY DESIGN:
Who Masked: Participant, Care Provider
Oversight: Data Monitoring Committee: Yes

ARMS (2):
- SMS-Web eAAP group (Experimental): electronic asthma action plan (eAAP) group
  Interventions: Other: electronic asthma action plan (eAAP)
- regular-care group (Active Comparator): written asthma action plan (WAAP) group
  Interventions: Other: written asthma action plan (WAAP)

INTERVENTIONS:
Other: electronic asthma action plan (eAAP) — An electronic asthma action plan (eAAP) will be provided to intervention group
  Arms: SMS-Web eAAP group
Other: written asthma action plan (WAAP) — A written asthma action plan will be given to control group arm
  Arms: regular-care group

SUMMARY:
Objectives:

The disease being studied is asthma. The main objective of this study is to assess the feasibility of the recruitment goals and also the logistical issues related to use of tele-health technology in developing electronic asthma action plan (eAAP) and communicate with asthma patients in a time period of 24 months. The goals are: 1) enable asthma patients to self-manage their asthma symptoms. The secondary, 2) help care providers to intervene appropriately based on the patient's health status. The secondary objective is to explore the cost-benefit and cost-effectiveness of the proposed technology. Our research group proposes to complete a feasibility study, with an interim analysis for a formal power calculation and then acquire ethics to report these results and study design with anticipated publication prior to proceeding with a full randomized controlled trial to assess the efficacy of this intervention. The outcome measure will be assessed and data will be presented in a 24-month time frame.

Aims and goals:

The main aim of our proposed study is to assist asthma patients to practice asthma self-management at home that will eventually enable them to control their asthma, and specifically, prevent asthma exacerbation. Therefore, the ultimate goal of our proposed study is to improve patient health outcome via enhancing patient-physician interaction and using a more practical asthma action plan model (eAAP) that could be followed easily by the patient and their doctor.

Our hypothesis is that asthma patients who have access to the electronic online action plan complimented by weekly text messages to reinforce adherence will have a reduced rate of asthma exacerbation. We further hypothesize that these subjects will have an improvement in secondary measures including quality of life, better asthma control and patient satisfaction. We also anticipate that such an approach in asthma management will be cost-effective as outlined below.

DETAILED DESCRIPTION:
In our study design we propose to use a web-based application and inform asthma patients through weekly Text Message (SMS) reminders to take their controller medication regularly and also a message to visit the web-based e-AAP and assess the current level of asthma control. This will be a two-way interaction and personalized feedback protocol to monitor patients at home and during daily activities. We will use an adequate sample size to provide an interim analysis of efficacy and the subsequent total number of subjects that will need to be enrolled. Each patient (in the relevant group, as explained below) will have his/her own profile, which will enable us to send and receive personalized (exchange) information using a web application process via cell phones. This approach will allow interaction between patient and asthma care counselor/ provider aiming to improve asthma control.

This study will test the hypothesis that using mobile phone reminder messages and web-based monitoring, as part of a structured care plan, will improve clinical outcomes; namely reduction in the rate of exacerbation, in patients with asthma. We also aim to explore the cost-effectiveness of this technology. Our research group proposes to complete a feasibility study, with an interim analysis for a formal power calculation and then acquire ethics to report these results and study design with anticipated publication prior to proceeding with a full randomized controlled trial to assess the efficacy of this intervention. We predict that using a combination of Internet and SMS messaging technology will empower patients to manage their asthma and eventually prevent asthma exacerbation based on their personalized action plan as well as a SMS application. We plan to compare the web-based/SMS reminder method with written action plan approach in a 24-month time frame, as explained later in this proposal.

ELIGIBILITY:
Inclusion Criteria:

1. Physician diagnosed asthma.
2. A history of an asthma exacerbation requiring oral corticosteroids or admission to Emergency Department/hospital in the previous year.
3. Ability to understand English and follow the material included in the two different interventions.
4. Ownership of a mobile phone with the capacity to support text messaging.
5. Patients on maintenance inhaled corticosteroids alone or with a combination inhaler. Subjects on other controller therapies will not be excluded as long as they fulfill these inclusion criteria.

   -

Exclusion Criteria:

1. Inability to provide written informed consent.
2. A history of smoking cigarettes for greater than ten pack years.
3. Not owning a mobile cell phone.
4. Subjects only taking a reliever medication and on no controller medication.
5. A history of significant co morbid disease judged by the investigator to preclude enrolment.
6. A history of an asthma exacerbation requiring oral corticosteroids in the previous six weeks.
7. Plans to move out of the study area in the next year. -

Ages: 19 Years to 85 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 100 (Actual)
Dates: Start 2014-08; Primary Completion 2017-06 (Estimated); Study Completion 2017-12 (Estimated)

PRIMARY OUTCOMES:
Reduction in the rate of asthma exacerbations | Number of asthma exacerbations will be assessed by Global Initiative for Asthma (GINA) standard assessment tool for 12 months post-intervention
  Tracking outcomes: All subjects will be asked to contact the study coordinator in the event of an asthma exacerbation. Subjects will also be seen at six and 12 months post intervention for the evaluation of health care utilization and record their asthma exacerbations. In addition, at this time baseline questionnaires will be repeated. They will also receive a telephone contact at three and nine months to document any recent exacerbations which they may have failed to call in with regard.

SECONDARY OUTCOMES:
the cost-effectiveness and cost-benefit of applying the SMS and web combination technology | Economic outcomes will be collected during the follow-up period (12 months after intervention). Cost-effectiveness will be assessed through decision-analytic modeling.
  Economic evaluation of health technologies is concerned with the trade-off between the incremental costs and incremental effectiveness of technologies and therefore requires collecting information on both costs and effectiveness at the individual level. The interventions in each arm of the trial are based on getting feedback from patients and as such substantial amount of information on the use of controller medications and asthma exacerbations will be collected. At month 6 and 12 after the intervention, participants will be invited to the study center for a detailed interview during which we will collect information on asthma-related resource use in the previous 6 months and will estimate participants' quality of life. As a surrogate for adherence, we will track prescriptions refills before and during the study using access to patient's PharmaNET data; which is feasible in BC, Canada.

CONTACTS AND LOCATIONS:
Overall Officials: Mark J FitzGerald, M.D., Principal Investigator — University of British Columbia
Locations (1):
- Centre for Clinical Epidemiology and Evaluation, Vancouver Coastal Health Research Institute, Vancouver, British Columbia, Canada

REFERENCES:
- See also: University of British Columbia Centre for Lung Health — http://www.centreforlunghealth.ca
- See also: Institute of Heart and Lung Health — http://heartandlung.ca/